CLINICAL TRIAL: NCT01559545
Title: A Randomized, Open Label, Active Control, Safety, Tolerability and Pharmacokinetics Study of Two Dr. Reddy's Formulations of Metronidazole Versus Immediate Release Metronidazole (Flagyl) in Patients With Mild to Moderate C. Difficile Associated Diarrhea (CDAD)
Brief Title: A Safety, Tolerability and Pharmacokinetic Study of Two Formulations of Metronidazole Versus Immediate Release Metronidazole in Patient With C. Difficile Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Collaborators: Reliance Clinical Research Services (Navi Mumbai, India) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFA-03-CD-002
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Clostridium Difficile Associated Diarrhea
Keywords: Clostridium difficile associated diarrhea; Metronidazole; CDAD
MeSH Terms: interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metronidazole (Active Comparator): Immediate release metronidazole
  Interventions: Drug: Metronidazole
- Metronidazole-DRF1 (Experimental): Modified release metronidazole (DRF1)
  Interventions: Drug: Metronidazole-DRF1
- Metronidazole-DRF2 (Experimental): Modified release metronidazole (DRF2)
  Interventions: Drug: Metronidazole-DRF2

INTERVENTIONS:
Drug: Metronidazole — Immediate release metronidazole 500 mg orally three times a day for 14 days
  Other Names: Flagyl®
  Arms: Metronidazole
Drug: Metronidazole-DRF1 — Modified release metronidazole (DRF1) 500 mg orally three times a day for 14 days.
  Other Names: Metronidazole
  Arms: Metronidazole-DRF1
Drug: Metronidazole-DRF2 — Modified release metronidazole (DRF2) 500 mg orally three times a day for 14 days.
  Other Names: Metronidazole
  Arms: Metronidazole-DRF2

SUMMARY:
Clostridium difficile bacteria can be a cause of significant diarrheal disease, particularly in people who have taken potent antibiotics. When C. difficile multiplies within the colon, it produces two toxins that cause inflammation and resultant abdominal pain, fever and diarrhea. Current treatment of mild to moderate disease is with immediate release metronidazole, an antibiotic that kills C. difficile. Dr. Reddy's Laboratories has developed a delayed release form of metronidazole to release just before the colon to increase the concentration of antibiotic in the colon to improve the effectiveness of metronidazole treatment and potentially to allow less whole body exposure to the antibiotic.

This study will measure the amount of metronidazole in the blood and stool of patients with C. difficile associated diarrhea (CDAD) to confirm that the new formulations are releasing the antibiotic as designed, immediately before the colon.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18 years of age or older
2. Mild to moderate C.difficile associated diarrhea (CDAD) with a positive stool C.difficile toxin (by ELISA).
3. Either a first episode of CDAD or a first recurrence (patients with more than 1 recurrence are not eligible)
4. Greater than 3 watery or unformed bowel movements in the prior 24 hours
5. Females of child bearing potential having a negative pregnancy test and taking adequate birth control measures.
6. Patients should not consume alcohol at least 12 hours prior to dosing (i.e. in-house monitoring) and until 48 hours after the last dose of drug administration (until Day 14).
7. Able to comprehend and give informed consent for the study and able to adhere to study schedules and protocol requirements.

Exclusion Criteria:

1. Known prior history of hypersensitivity to metronidazole or other nitroimidazole derivatives
2. Life expectancy ≤ 60 days
3. Sepsis, severe sepsis, or septic shock
4. Signs or symptoms of peritonitis, megacolon or ileus
5. History of ulcerative colitis or Crohn's disease
6. Oral or parenteral antibiotic therapy with metronidazole or vancomycin or other drugs effective in treating DCAD (e.g., bacitracin, fusidic acid) within the 1 week prior to enrollment
7. Recent history of significant drug or alcohol abuse within 1 year
8. Any findings on physical examination, medical history, 12-lead ECG or clinical laboratory tests which, in the judgment of the Principal Investigator, would exclude patients from participating in the study
9. Patients with history of blood dyscrasias, porphyria and active non-infectious disease of the central nervous system
10. Patients with history of rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
11. Pregnant or lactating female patients
12. Participation within 30 days before the start of this study in any experimental drug or device study, or currently participating in a study in which the administration of investigational drug or device within 60 days is anticipated
13. Unable to participate in the study for any reason in the opinion of the Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Tolerability | 44 Days
  Tolerability as assessed by physical examination, ECG, clinical laboratory tests and adverse events
Pharmacokinetics | 14 Days
  Systemic pharmacokinetics of metronidazole on Days 1 and 14. Intraluminal colonic concentration of metronidazole as reflected in excreted stool on Days 1 and 14.

SECONDARY OUTCOMES:
Clinical Cure | 44 Days
  Response rate to treatment 2 days after completion of 14 days of metronidazole treatment with no recurrence 30 days after 14 days of metronidazole treatment (Day 44).
Recurrence Rate | 44 Days
  Recurrence defined as re-establishment of diarrhea after clinical cure.
30-Day Cure Rate | 44 Days
  Clinical cure with no recurrence and no retreatment for 30 days after 14 days of metronidazole treatment (Day 44).

CONTACTS AND LOCATIONS:
Overall Officials: Dilip Pawar, MD, Study Director — Dr. Reddy's Laboratories Limited
Locations (12):
- India (12):
  - Dr. B.R. Ambedkar Medical College, Bangalore, Karnataka
  - St. John's Medical College and Hospital, Bangalore, Karnataka
  - PRS Hospitals, Trivandrum, Kerala
  - B.Y.L. Nair Hospital, Mumbai, Maharashtra
  - Chopda Research and Medical Center Pvt, Nashik, Maharashtra
  - Deenanath Mangeshkar Hospital, Pune, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - S.P. Medical College and Hospital, Bikaner, Rajasthan
  - Apex Medicical College, Jaipur, Rajasthan
  - Meenakshi Mission Hospital and Research Center, Madurai, Tamil Nadu
  - SKS Hospital India Pvt. Ltd., Salem, Tamil Nadu
  - Heritage Hospital, Lanka, Varanasi